CLINICAL TRIAL: NCT01813201
Title: A Randomized and Double-blind Study to Evaluate the Benefit of the Treatment With Testosterone in Chronic Heart Failure Testosterone Deficiency Subjects
Brief Title: Benefit of the Treatment With Testosterone in Chronic Heart Failure Testosterone Deficiency Subjects
Acronym: TIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TIC-0911; 2009-016498-13 (EudraCT Number)
Record Dates: First submitted 2011-06-22; First posted 2013-03-18 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2014-11

CONDITIONS: Heart Failure
Keywords: Testosterone; Anabolic deterioration
MeSH Terms: conditions — Heart Failure | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone undecanoate (Active Comparator): Testosterone undecanoate intramuscular long-acting, 1000 mg/dose, administered at inclusion and every 12 weeks for 9 months (4 dose)
  Interventions: Drug: Testosterone undecanoate
- Saline isotonic solution (Placebo) (Placebo Comparator): Placebo (saline isotonic solution)administered at inclusion and every 12 weeks for 9 months (4 dose) (control group).
  Interventions: Drug: Saline isotonic solution

INTERVENTIONS:
Drug: Testosterone undecanoate — Testosterone undecanoate intramuscular long-acting, 1000 mg/dose, administered at inclusion and every 12 weeks for 9 months (4 dose) (testosterone group) against the administration of placebo (saline isotonic solution).
  Other Names: Reandron®
  Arms: Testosterone undecanoate
Drug: Saline isotonic solution — Saline isotonic solution (placebo)intramuscular,administered at inclusion and every 12 weeks for 9 months (4 dose)
  Arms: Saline isotonic solution (Placebo)

SUMMARY:
The purpose of this clinical trial is to determine whether intermittent administration of testosterone against placebo is associated with a reduction of mortality and heart failure hospitalizations at 1 year, in male patients with advanced heart failure and testosterone deficiency.

DETAILED DESCRIPTION:
Heart Failure (HF) represents one of the major social and health problems, for its high prevalence and its huge economic impact, as well as the elevated morbidity and mortality associated. In Spain, the estimated prevalence is 7% over 45 years old, and it increases until 18% over 75 years old. Currently, HF is the leading cause of hospital admission over 65 years and the mortality for patients with symptomatic HF remains worse than the majority of cancers. The estimated minimum expenditure is 1.1% of total health care costs and 2% of specialized medical care. This accounts for a staggeringly large financial burden on the health care system.

Chronic HF is a complex disease, whose progression involves multiple pathophysiological systems. It is well established the deleterious effect of activation of renin-angiotensin-aldosterone and sympathetic nervous systems. The blockage of these systems by beta-blockers, angiotensin converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARBs) and aldosterone antagonists has improved prognosis. However, in spite of these therapies, the prognosis of patients with chronic HF remains poor.

During the HF progression to advanced stages, it has been shown an anabolic and metabolic deterioration, resulting in a predominance of catabolic processes. The deficiency of anabolic hormones correlates with greater severity of symptoms, activation of neuroendocrine and inflammatory systems, insulin resistance, metabolic impairment, exercise intolerance, anemia and cardiac cachexia. All these processes take part of the final progression of the HF disease until death, when HF becomes a systemic disease. In men with HF, levels of testosterone (the main anabolic hormone) are decreased; in fact, 30% of men have levels below the 10th percentile of a reference healthy population adjusted for age. The deterioration of anabolic hormones correlates inversely with the severity of HF disease and it determines a higher mortality. In fact, low testosterone levels are associated with reduced cardiac output, greater symptomatic limitation and higher mortality. Therefore, testosterone deficiency in men with HF has a detrimental impact on symptoms and prognosis.

In addition, testosterone has shown to have beneficial effects on HF patients, such as vasodilatation of coronary and peripheral arteries, inotropic effects, reduction of neurohormonal activation, anti-inflammatory and immunomodulatory actions, reduction of cytokine production and improvement of muscle strength. All these actions have a potential benefit in patients with HF, because they are involved in the progression of the disease, especially at advanced stages.

The rational approach "testosterone replacement for improving the prognosis of patients with advanced HF and testosterone deficiency" has strong pathophysiological plausibility. To date, no other clinical trials have evaluated the effect of testosterone replacement on morbidity and mortality.

However, in the last years, numerous editorials in leading journals have concluded on the need to clarify the effect of testosterone therapy on cardiac function and the morbimortality in patients with advanced HF.

Our group has worked in the last years in this field, confirming the presence of a testosterone deficiency in men with chronic HF, which is associated with a worse prognosis and a greater decline in exercise capacity.

Therefore, the investigators propose a clinical trial of morbimortality in a population with advanced heart failure and associated deficiency on testosterone; in which, the previous background justifies the potential benefit of testosterone replacement therapy. In addition, the large clinical impact of this disease supports the priority need of an independent study.

ELIGIBILITY:
Inclusion Criteria:

* At least one hospital admission for HF.
* Stable clinical status, New York Heart Association (NYHA) functional class II-IV.
* Left ventricular ejection fraction of less than 40%
* NT-proBNP concentration greater than 1000 pg / ml.
* Total testosterone and free testosterone deficiency measured in the last month
* Age >18 years.
* Patients who have given their written informed consent.

Exclusion Criteria:

* No informed consent.
* Taking oral anticoagulants
* Severe valvular heart disease with an indication for surgical repair.
* Extracardiac disease with an estimated prognosis of less than 1 year.
* History of androgen-dependent prostate cancer, benign prostate hyperplasia treatment or prostate-specific antigen (PSA)> 3 ng / ml.
* History of breast carcinoma or liver tumor
* Severe renal impairment (glomerular filtration rate <30 ml / kg / min).
* Acute coronary syndrome in the last year
* Renal or hepatic failure
* Uncontrolled hypertension
* Erythrocytosis (hematocrit> 5%)
* Hypersensitivity to testosterone or any excipients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Death | 1 year
  Death from any cause or hospitalization for heart failure or decompensation of heart failure requiring intravenous drug for stabilization.

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality from cardiovascular causes, for HF and other causes.
Hospital readmissions for any reason. | 1 year
Number of decompensated heart failure who have required intravenous medication for stabilization. | 1 year
Changes in test quality of life (Minnesota Living Heart Failure) and clinical modified Framingham score. | 1 year
Changes in cardiac function parameters assessed by echocardiography and natriuretic peptide (NT)-proBNP concentration. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Domingo A Pascual-Figal, MD, PhD, Principal Investigator — Hospital Universitario Virgen Arrixaca; Antoni Bayes-Genis, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Cardiology Service, Hospital Universitario Virgen de la Arrixaca, Murcia, Spain

REFERENCES:
- [Background] Rodriguez-Artalejo F, Banegas Banegas JR, Guallar-Castillon P. [Epidemiology of heart failure]. Rev Esp Cardiol. 2004 Feb;57(2):163-70. Spanish. PMID 14967113
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Pugh PJ, English KM, Jones TH, Channer KS. Testosterone: a natural tonic for the failing heart? QJM. 2000 Oct;93(10):689-94. doi: 10.1093/qjmed/93.10.689. No abstract available. PMID 11029481
- [Background] Malkin C, Jones T, Channer K. Testosterone in chronic heart failure. Front Horm Res. 2009;37:183-196. doi: 10.1159/000176053. PMID 19011297
- [Background] Pugh PJ, Jones RD, Jones TH, Channer KS. Heart failure as an inflammatory condition: potential role for androgens as immune modulators. Eur J Heart Fail. 2002 Dec;4(6):673-80. doi: 10.1016/s1388-9842(02)00162-9. PMID 12453536
- [Background] Anker SD, Al-Nasser FO. Chronic heart failure as a metabolic disorder. Heart Fail Monit. 2000;1(2):42-9. PMID 12634873
- [Background] Anker SD, Chua TP, Ponikowski P, Harrington D, Swan JW, Kox WJ, Poole-Wilson PA, Coats AJ. Hormonal changes and catabolic/anabolic imbalance in chronic heart failure and their importance for cardiac cachexia. Circulation. 1997 Jul 15;96(2):526-34. doi: 10.1161/01.cir.96.2.526. PMID 9244221
- [Background] Kontoleon PE, Anastasiou-Nana MI, Papapetrou PD, Alexopoulos G, Ktenas V, Rapti AC, Tsagalou EP, Nanas JN. Hormonal profile in patients with congestive heart failure. Int J Cardiol. 2003 Feb;87(2-3):179-83. doi: 10.1016/s0167-5273(02)00212-7. PMID 12559538
- [Background] Moriyama Y, Yasue H, Yoshimura M, Mizuno Y, Nishiyama K, Tsunoda R, Kawano H, Kugiyama K, Ogawa H, Saito Y, Nakao K. The plasma levels of dehydroepiandrosterone sulfate are decreased in patients with chronic heart failure in proportion to the severity. J Clin Endocrinol Metab. 2000 May;85(5):1834-40. doi: 10.1210/jcem.85.5.6568. PMID 10843161
- [Background] Jankowska EA, Biel B, Majda J, Szklarska A, Lopuszanska M, Medras M, Anker SD, Banasiak W, Poole-Wilson PA, Ponikowski P. Anabolic deficiency in men with chronic heart failure: prevalence and detrimental impact on survival. Circulation. 2006 Oct 24;114(17):1829-37. doi: 10.1161/CIRCULATIONAHA.106.649426. Epub 2006 Oct 9. PMID 17030678
- [Background] Jankowska EA, Filippatos G, Ponikowska B, Borodulin-Nadzieja L, Anker SD, Banasiak W, Poole-Wilson PA, Ponikowski P. Reduction in circulating testosterone relates to exercise capacity in men with chronic heart failure. J Card Fail. 2009 Jun;15(5):442-50. doi: 10.1016/j.cardfail.2008.12.011. Epub 2009 Feb 10. PMID 19477405
- [Background] P Peñafiel, DA Pascual, B. Redondo, P Nicolas, PL Tornel, J Sanchez-Mas, G de la Morena, M Valdés. Anabolic deficiency as determinant of functional impairment and prognosis in heart failure patients. European journal of Heart Failure 2007;6(supl 1):146.
- [Background] Pugh PJ, Jones TH, Channer KS. Acute haemodynamic effects of testosterone in men with chronic heart failure. Eur Heart J. 2003 May;24(10):909-15. doi: 10.1016/s0195-668x(03)00083-6. PMID 12714022
- [Background] Malkin CJ, Jones TH, Channer KS. The effect of testosterone on insulin sensitivity in men with heart failure. Eur J Heart Fail. 2007 Jan;9(1):44-50. doi: 10.1016/j.ejheart.2006.04.006. Epub 2006 Jul 7. PMID 16828341
- [Background] Rauchhaus M, Doehner W, Anker SD. Heart failure therapy: testosterone replacement and its implications. Eur Heart J. 2006 Jan;27(1):10-2. doi: 10.1093/eurheartj/ehi653. Epub 2005 Nov 16. No abstract available. PMID 16291772
- [Background] Pugh PJ, Jones RD, West JN, Jones TH, Channer KS. Testosterone treatment for men with chronic heart failure. Heart. 2004 Apr;90(4):446-7. doi: 10.1136/hrt.2003.014639. No abstract available. PMID 15020527
- [Background] Malkin CJ, Pugh PJ, West JN, van Beek EJ, Jones TH, Channer KS. Testosterone therapy in men with moderate severity heart failure: a double-blind randomized placebo controlled trial. Eur Heart J. 2006 Jan;27(1):57-64. doi: 10.1093/eurheartj/ehi443. Epub 2005 Aug 10. PMID 16093267
- [Background] Caminiti G, Volterrani M, Iellamo F, Marazzi G, Massaro R, Miceli M, Mammi C, Piepoli M, Fini M, Rosano GM. Effect of long-acting testosterone treatment on functional exercise capacity, skeletal muscle performance, insulin resistance, and baroreflex sensitivity in elderly patients with chronic heart failure a double-blind, placebo-controlled, randomized study. J Am Coll Cardiol. 2009 Sep 1;54(10):919-27. doi: 10.1016/j.jacc.2009.04.078. PMID 19712802
- [Background] Aukrust P, Ueland T, Gullestad L, Yndestad A. Testosterone: a novel therapeutic approach in chronic heart failure? J Am Coll Cardiol. 2009 Sep 1;54(10):928-9. doi: 10.1016/j.jacc.2009.05.039. No abstract available. PMID 19712803
- [Background] Pascual-Figal DA, Tornel PL, Valdes M. Letter by Pascual-Figal et al regarding article, "Anabolic deficiency in men with chronic heart failure: prevalence and detrimental impact on survival". Circulation. 2007 May 29;115(21):e548; author reply e549. doi: 10.1161/CIRCULATIONAHA.106.685040. No abstract available. PMID 17533191
- [Derived] Navarro-Penalver M, Perez-Martinez MT, Gomez-Bueno M, Garcia-Pavia P, Lupon-Roses J, Roig-Minguell E, Comin-Colet J, Bayes-Genis A, Noguera JA, Pascual-Figal DA. Testosterone Replacement Therapy in Deficient Patients With Chronic Heart Failure: A Randomized Double-Blind Controlled Pilot Study. J Cardiovasc Pharmacol Ther. 2018 Nov;23(6):543-550. doi: 10.1177/1074248418784020. Epub 2018 Jun 21. PMID 29929385
- See also: MeSH Terms — http://www.ncbi.nlm.nih.gov/mesh/68006333
- See also: Spanish Cardiology Society — http://www.secardiologia.es/